CLINICAL TRIAL: NCT00163293
Title: Effect of Low Dose Continuous Treatment With Ciclesonide Over One Year on the Time to First Exacerbation in Children With Mild Asthma Versus Intermittent Treatment for Exacerbations
Brief Title: Efficacy of Ciclesonide Inhaled Once Daily Versus Other Corticosteroids Used for Treatment of Mild Asthma in Children (4 to 11 Years) (BY9010/CA-101)
Acronym: POPCICLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/CA-101; 2007-003736-34 (EudraCT Number); U1111-1189-7814 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Exacerbation
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ciclesonide 100 µg (Active Comparator): Ciclesonide 100 µg, metered-dose inhaler, two puffs once daily, in the evening, for up to 12 months.
  Interventions: Drug: Ciclesonide
- Ciclesonide 200 µg (Active Comparator): Ciclesonide 200 µg, metered-dose inhaler, two puffs once daily, in the evening, for up to 12 months.
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide — Ciclesonide metered-dose inhaler
  Other Names: Alvesco®
  Arms: Ciclesonide 100 µg; Ciclesonide 200 µg
Drug: Placebo — Ciclesonide placebo-matching metered-dose inhaler
  Arms: Placebo

SUMMARY:
The aim of this study is to compare the efficacy of ciclesonide with respect to reduction of the number of asthma exacerbations in children with mild persistent asthma. Treatment medication will be administered as follows: ciclesonide will be inhaled once daily, using one of the two dose levels versus placebo together with other corticosteroids used as intermittent treatment. The study duration consists of a baseline period (3 to 4 weeks) and a treatment period (12 months). The study will provide further data on safety and tolerability of ciclesonide.

DETAILED DESCRIPTION:
The drug being tested in this study is called ciclesonide. Ciclesonide is being tested to treat children who have mild asthma.

The study enrolled 240 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Ciclesonide 100 µg
* Ciclesonide 200 µg
* Placebo (dummy inactive inhalation) - this is a metered-dose inhaler that looks like the study drug but has no active ingredient.

All participants were asked to take two puffs from a metered-dose inhaler once daily, in the evening, for up to 12 months.

This multi-center trial was conducted in Canada, Hungary and South Africa. The overall time to participate in this study was 12 months preceded by a baseline washout period of 3 to 4 weeks. Participants made multiple visits to the clinic including a safety follow-up visit within 30 days of the last treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Outpatients
* Symptoms consistent with the diagnosis of asthma for at least 12 months
* Forced Expiratory Volume in one Second (FEV) at least 80% of predicted
* Participants who have a history of reversible airway obstruction
* Good health with the exception of asthma

Main Exclusion Criteria:

* History of life-threatening asthma
* A hospitalization for asthma within the last 3 months, or more than two hospitalizations for asthma within the last year
* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Participants suffering from relevant lung diseases causing alternating impairment in lung function (e.g. chronic bronchitis or emphysema)
* Prematurely born children (<36 weeks of gestation)
* Smokers
* Pregnancy (or intention to become pregnant during the course of the trial), breast feeding or lack of safe contraception by female of child-bearing potential

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (7):
- Canada (5):
  - Altana Pharma/Nycomed, Calgary
  - Altana Pharma/Nycomed, Fleurimont
  - Altana Pharma/Nycomed, London
  - Altana Pharma/Nycomed, London,ON
  - Altana Pharma/Nycomed, Winnipeg
- Altana Pharma/Nycomed, Budapest, Hungary
- Altana Pharma/Nycomed, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in Canada, Hungary and South Africa from 24 January 2005 to 25 June 2009.
Pre-assignment Details: Children who experienced symptoms consistent with mild asthma for at least 12 months were enrolled in 1 of 3 treatment groups: once a day placebo, 100 µg or 200 µg ciclesonide.
Groups:
- Placebo: Ciclesonide placebo-matching, metered-dose inhaler, two puffs once daily, in the evening, for up to 12 months.
Period: Overall Study
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Started | 79 | 76 | 85
Completed | 66 | 69 | 66
Not Completed | 13 | 7 | 19

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo | Total
Number analyzed (Participants) | 79 | 76 | 84 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (2.06) | 7.7 (1.84) | 8.1 (2.19) | 7.9 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 34 | 98
  Male | 46 | 45 | 50 | 141
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 6 | 6 | 18
  Black | 4 | 2 | 5 | 11
  Caucasian | 55 | 53 | 59 | 167
  Other | 14 | 15 | 14 | 43
Weight [Mean (Standard Deviation); unit: kg] — Weight data was only available for n=77, 76, 84 participants, respectively.
  kg | 29.90 (9.701) | 30.01 (9.247) | 33.13 (11.640) | 31.08 (10.365)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data was only available for n=77, 76, 84 participants, respectively.
  kg/m^2 | 17.30 (3.107) | 17.69 (2.977) | 18.68 (4.069) | 17.91 (3.478)
Smoking Classification (Non-smoker) [Number; unit: participants] | 79 | 76 | 84 | 239

OUTCOME MEASURES:

1. Primary Outcome: Time to First Asthma Exacerbation
Description: Time to first asthma exacerbation is defined as the time in days until the first asthma exacerbation, or to the end of treatment visit. In the absence of an exacerbation, an early treatment discontinuation is treated as a censored observation on the day following the last use of study drug.
Time Frame: Up to 12 months
Population: Intention to Treat (ITT) analysis set included all participants of the full analysis set who received at least one dose of study medication and had at least one post-baseline measurement of the primary efficacy outcome.
Measure: Mean (Standard Error); unit: days
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
days | 225.1 (14.73) | 249.5 (14.79) | 227.2 (15.20)
Statistical Analysis 1: Comparison: Ciclesonide 100 µg vs Placebo; Test type: Superiority or Other; p = 0.6625, Log Rank
Statistical Analysis 2: Comparison: Ciclesonide 200 µg vs Placebo; Test type: Superiority or Other; p = 0.7303, Log Rank

2. Primary Outcome: Exacerbations (Post-hoc Analysis of Annual Rates)
Description: A model-based analysis of asthma exacerbation was performed to adjust to important covariables. The distribution of the data suggested a Poisson regression modeling (zero inflated) strategy. After a variable selection process considering also variable-by-treatment interactions, the variables centre, age [years] and race were identified to be important beside treatment. The parameters centre and age [years] were allocated to zero-model part and the variables treatment and race to the Poisson model part. The estimates of the per-treatment rates are based on a negative-binomial distribution.
Time Frame: Up to 12 months
Population: ITT analysis set included all participants of the full analysis set who received at least one dose of study medication and had at least one post-baseline measurement of the primary efficacy outcome.
Measure: Least Squares Mean (Standard Error); unit: number of events per year
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
number of events per year | 0.9343 (0.2909) | 0.8794 (0.2747) | 1.2621 (0.2768)
Statistical Analysis 1: Comparison: Ciclesonide 100 µg vs Placebo; Test type: Superiority or Other; p = 0.1291, Wald Chi-square; zero inflated Poisson model: adjustment for centre and age [yrs] (zero model), treatment and race (Poisson model)
Statistical Analysis 2: Comparison: Ciclesonide 200 µg vs Placebo; Test type: Superiority or Other; p = 0.0145, Wald Chi-square; zero inflated Poisson model: adjustment for centre and age [yrs] (zero model), treatment and race (Poisson model)

3. Secondary Outcome: Growth Velocity as Assessed by Stadiometric Height Measurement
Description: Standing height measured in millimeters (mm) with a wall-mounted stadiometer.
Time Frame: Up to 12 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
mm/year | 55.32 (25.81) | 64.60 (27.31) | 54.91 (21.78)

4. Secondary Outcome: Mean Rate of Asthma Exacerbations Per Year
Description: Rate of asthma exacerbations per year is equal to total number of asthma exacerbations during treatment/time on treatment (year).
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of exacerbations per year
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
number of exacerbations per year | 0.88 (1.366) | 0.85 (1.310) | 3.28 (19.874)
Statistical Analysis 1: Comparison: Ciclesonide 100 µg vs Placebo; Test type: Superiority or Other; p = 0.4754, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ciclesonide 200 µg vs Placebo; Test type: Superiority or Other; p = 0.6844, Kruskal-Wallis

5. Secondary Outcome: Duration of Exacerbations
Description: Duration of exacerbation was defined as the time in days when the criteria for an exacerbation were met to the time when peak flow measurements returned to baseline.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
days | 9.17 (6.198) | 9.31 (7.650) | 7.92 (4.061)

6. Secondary Outcome: Number of Exacerbations Per Participant
Description: The mean number of asthma exacerbations per participant is reported.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: exacerbations
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
exacerbations | 0.72 (1.025) | 0.78 (1.028) | 0.95 (1.316)

7. Secondary Outcome: Percentage of Participants Who Dropped-out Due to Asthma Exacerbation
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percentage of participants | 1.3 | 1.3 | 4.8

8. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) (Absolute Value)
Description: FEV1 is the maximal amount of air forcefully exhaled from the lungs in one second. Spirometry was used for assessment of FEV1. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Months 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants of the full analysis set who received at least one dose of study medication and had at least one post-baseline measurement of the primary efficacy outcome. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
liters
  Change at Month 1 (n=78, 76, 81) | 0.019 (0.1715) | 0.018 (0.1639) | 0.012 (0.1627)
  Change at Month 2 (n=76, 73, 77) | 0.024 (0.1416) | 0.060 (0.1582) | 0.005 (0.1416)
  Change at Month 4 (n=68, 72, 75) | 0.065 (0.1483) | 0.083 (0.1486) | 0.076 (0.1725)
  Change at Month 6 (n=67, 72, 72) | 0.091 (0.1714) | 0.125 (0.1975) | 0.078 (0.1855)
  Change at Month 8 (n=66, 71, 68) | 0.075 (0.2144) | 0.126 (0.2089) | 0.120 (0.1855)
  Change at Month 10 (n=66, 69, 67) | 0.143 (0.1458) | 0.168 (0.1910) | 0.146 (0.1609)
  Change at Month 12 (n=65, 69, 65) | 0.161 (0.2022) | 0.185 (0.2024) | 0.178 (0.1593)

9. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) (Percent Predicted)
Description: as for outcome 8
Time Frame: Baseline and Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percent predicted FEV1
  Change at Month 1 (n=78, 76, 81) | 1.0 (10.96) | 0.6 (9.67) | 1.0 (9.06)
  Change at Month 2 (n=76, 73, 77) | 1.4 (8.50) | 3.4 (9.60) | 0.3 (8.05)
  Change at Month 4 (n=68, 72, 75) | 4.0 (8.69) | 4.6 (9.31) | 5.1 (9.83)
  Change at Month 6 (n=67, 72, 72) | 5.5 (10.00) | 7.2 (11.35) | 4.9 (10.93)
  Change at Month 8 (n=66, 71, 68) | 4.4 (12.44) | 6.5 (12.25) | 7.1 (10.24)
  Change at Month 10 (n=66, 69, 67) | 8.6 (9.41) | 9.1 (10.48) | 8.7 (9.22)
  Change at Month 12 (n=65, 69, 65) | 9.5 (10.96) | 10.1 (11.29) | 10.4 (9.89)

10. Secondary Outcome: Morning and Evening Peak Expiratory Flow (PEF) Measurements by Diary Entries
Description: PEF is the maximum speed of expiration. Spirometry was used for assessment of PEF.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
liters/second
  Month 1, Evening PEF (n=78, 76, 80) | 235.72 (63.882) | 238.16 (52.565) | 241.89 (70.619)
  Month 1, Morning PEF (n=78, 76, 81) | 232.09 (64.933) | 234.41 (52.908) | 233.81 (66.039)
  Month 2, Evening PEF (n=76, 71, 77) | 241.07 (58.604) | 241.16 (50.422) | 244.67 (67.846)
  Month 2, Morning PEF (n=76, 72, 77) | 236.92 (61.243) | 236.42 (52.323) | 239.07 (70.132)
  Month 4, Evening PEF (n=68, 72, 75) | 249.75 (58.528) | 243.52 (49.076) | 245.91 (65.802)
  Month 4, Morning PEF (n=68, 71, 76) | 242.93 (56.658) | 241.91 (48.498) | 240.16 (65.211)
  Month 6, Evening PEF (n=67, 72, 73) | 251.88 (60.255) | 249.36 (59.294) | 246.44 (63.946)
  Month 6, Morning PEF (n=67, 72, 73) | 246.44 (59.781) | 246.75 (60.020) | 238.81 (63.419)
  Month 8, Evening PEF (n=66, 70, 69) | 253.49 (59.666) | 250.92 (51.376) | 245.72 (61.399)
  Month 8, Morning PEF (n=66, 71, 69) | 247.24 (59.806) | 246.97 (51.592) | 239.73 (61.733)
  Month 10, Evening PEF (n=65, 70, 68) | 254.21 (56.815) | 256.44 (56.469) | 251.69 (60.704)
  Month 10, Morning PEF (n=66, 70, 68) | 247.94 (60.418) | 254.04 (56.719) | 246.23 (62.805)
  Month 12, Evening PEF (n=68, 71, 70) | 255.97 (57.291) | 263.87 (58.469) | 261.88 (61.383)
  Month 12, Morning PEF (n=75, 73, 78) | 245.84 (59.834) | 258.62 (57.009) | 250.55 (63.204)

11. Secondary Outcome: Change From Baseline in PEF by Diary Entries
Description: PEF is the maximum speed of expiration. Spirometry was used for assessment of PEF. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
liters/second
  Change at Month 1, Evening PEF (n=78, 76, 80) | 8.46 (17.952) | 8.54 (19.474) | 6.06 (39.183)
  Change at Month 1, Morning PEF (n=78, 76, 81) | 11.69 (21.268) | 10.82 (20.372) | 7.54 (25.697)
  Change at Month 2, Evening PEF (n=76, 71, 77) | 13.66 (28.491) | 13.04 (20.890) | 10.83 (40.563)
  Change at Month 2, Morning PEF (n=76, 72, 77) | 17.12 (32.068) | 14.30 (22.649) | 14.29 (37.228)
  Change at Month 4, Evening PEF (n=68, 72, 75) | 20.41 (22.058) | 16.01 (21.547) | 13.62 (37.990)
  Change at Month 4, Morning PEF (n=68, 71, 76) | 21.33 (26.603) | 18.24 (22.808) | 16.28 (34.841)
  Change at Month 6, Evening PEF (n=67, 72, 73) | 22.44 (28.236) | 21.86 (38.280) | 13.14 (33.321)
  Change at Month 6, Morning PEF (n=67, 72, 73) | 24.82 (30.613) | 24.68 (40.981) | 14.44 (29.950)
  Change at Month 8, Evening PEF (n=66, 70, 69) | 25.47 (27.430) | 21.38 (28.648) | 13.30 (37.061)
  Change at Month 8, Morning PEF (n=66, 71, 69) | 27.16 (32.530) | 23.76 (29.089) | 16.03 (34.017)
  Change at Month 10, Evening PEF (n=65, 70, 68) | 25.68 (30.945) | 26.78 (34.255) | 18.04 (38.209)
  Change at Month 10, Morning PEF (n=66, 70, 68) | 27.86 (38.406) | 29.84 (36.390) | 21.25 (34.940)
  Change at Month 12, Evening PEF (n=68, 71, 70) | 28.24 (28.811) | 33.35 (38.772) | 25.38 (43.284)
  Change at Month 12, Morning PEF (n=75, 73, 78) | 26.84 (32.932) | 34.31 (41.166) | 24.37 (39.312)

12. Secondary Outcome: Change From Baseline in Diurnal PEF Fluctuation
Description: Diurnal PEF Fluctuation is equal to [(Higher PEF - Lower PEF)/0.5*(Higher PEF + Lower PEF)] * 100%. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent fluctuation
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percent fluctuation
  Change at Month 1 (n=78, 76, 80) | -0.59 (3.970) | 0.06 (3.772) | 0.00 (3.867)
  Change at Month 2 (n=76, 71, 77) | -0.13 (5.009) | -0.16 (4.131) | 0.15 (5.084)
  Change at Month 4 (n=68, 71, 75) | -0.65 (5.251) | -1.01 (3.784) | -0.55 (4.421)
  Change at Month 6 (n=67, 72, 73) | -1.01 (4.351) | -0.22 (5.860) | -0.47 (4.280)
  Change at Month 8 (n=66, 70, 69) | -1.12 (4.830) | -1.21 (3.757) | -1.11 (4.048)
  Change at Month 10 (n=64, 70, 68) | -1.46 (5.221) | -0.70 (4.319) | -1.14 (4.059)
  Change at Month 12 (n=68, 70, 70) | -1.81 (4.913) | -0.62 (4.440) | -1.26 (4.187)

13. Secondary Outcome: Total Asthma Symptom Score by Diary Entries
Description: Total Asthma Score = daytime asthma score + night-time asthma score, where higher score indicates worsening of disease. Night-time asthma score is assessed on a 5 point scale where 0=No symptoms, slept through the night, 1=Slept well but some complaints in the morning, 2=Woke up once because of asthma (including early wakening), 3=Woke up several times because of asthma (including early wakening) and 4=Bad night, awake most of the night because of asthma. Day-time asthma score is assessed on a 5 point scale where 0= Very well, no symptoms, 1= One episode of wheezing, cough or breathlessness, 2= More than one episode of wheezing, cough or breathlessness without interfering with normal activities, 3= Wheezing, cough or shortness of breath most of the day which interfered to some extent with normal activities and 4= Asthma very bad. Unable to carry out daily activities as usual.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
score on a scale
  Month 1 (n=77, 75, 79) | 0.37 (0.489) | 0.22 (0.329) | 0.32 (0.535)
  Month 2 (n=76, 70, 77) | 0.26 (0.424) | 0.14 (0.246) | 0.28 (0.484)
  Month 4 (n=68, 72, 75) | 0.18 (0.342) | 0.12 (0.178) | 0.24 (0.359)
  Month 6 (n=67, 72, 73) | 0.16 (0.289) | 0.17 (0.294) | 0.18 (0.289)
  Month 8 (n=66, 69, 69) | 0.17 (0.283) | 0.13 (0.243) | 0.23 (0.414)
  Month 10 (n=64, 70, 68) | 0.12 (0.253) | 0.11 (0.227) | 0.24 (0.490)
  Month 12 (n=68, 69, 70) | 0.11 (0.240) | 0.08 (0.129) | 0.15 (0.338)

14. Secondary Outcome: Percentage of Nights With Nocturnal Awakenings Due to Asthma Symptoms
Description: Nocturnal awakenings due to asthma symptoms were recorded in the participant's diary.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of nights
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percentage of nights
  Month 1 (n=78, 75, 80) | 2.40 (6.159) | 1.64 (4.256) | 1.85 (4.223)
  Month 2 (n=76, 73, 77) | 1.96 (5.877) | 0.62 (2.364) | 1.73 (4.662)
  Month 4 (n=68, 72, 75) | 1.33 (4.017) | 0.86 (2.139) | 1.54 (4.106)
  Month 6 (n=67, 72, 73) | 0.87 (2.527) | 1.51 (3.288) | 1.26 (3.235)
  Month 8 (n=66, 70, 69) | 1.62 (4.129) | 1.05 (2.823) | 1.82 (5.024)
  Month 10 (n=66, 70, 68) | 1.93 (7.106) | 0.59 (2.220) | 1.88 (5.468)
  Month 12 (n=74, 73, 78) | 0.41 (1.554) | 1.84 (11.769) | 0.53 (1.853)

15. Secondary Outcome: Rescue Medication Use Per Day
Description: Salbutamol (100 μg/puff) was used as rescue medication according to the individual needs of the participant. Each use was documented in the participant's diary.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: puffs/day
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
puffs/day
  Month 1 (n=57, 51, 54) | 1.00 (1.345) | 0.83 (1.148) | 0.87 (0.910)
  Month 2 (n=53, 40, 46) | 0.99 (1.296) | 0.53 (0.728) | 0.97 (1.298)
  Month 4 (n=48, 47, 51) | 0.88 (1.300) | 1.18 (1.595) | 1.27 (1.984)
  Month 6 (n=45, 43, 44) | 0.79 (1.084) | 1.07 (1.329) | 0.92 (1.583)
  Month 8 (n=38, 42, 45) | 1.01 (1.530) | 1.13 (1.950) | 0.97 (1.219)
  Month 10 (n=38, 41, 39) | 0.93 (1.423) | 0.95 (1.243) | 0.83 (1.113)
  Month 12 (n=36, 40, 40) | 0.71 (0.897) | 1.01 (1.360) | 0.75 (1.152)

16. Secondary Outcome: Percentage of Rescue Medication Free Days
Description: Days without use of rescue medication documented in the participant's diary were reported.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percentage of days
  Month 1 (n=55, 53, 54) | 47.94 (44.405) | 47.34 (44.984) | 44.37 (45.367)
  Month 2 (n=52, 41, 48) | 48.78 (46.442) | 54.46 (46.668) | 45.31 (47.761)
  Month 4 (n=49, 48, 52) | 49.91 (48.274) | 46.51 (45.209) | 45.91 (46.328)
  Month 6 (n=47, 44, 45) | 49.63 (48.084) | 48.14 (45.321) | 49.42 (47.515)
  Month 8 (n=39, 42, 44) | 47.93 (45.170) | 50.50 (46.100) | 45.22 (45.002)
  Month 10 (n=40, 40, 37) | 46.22 (47.901) | 49.78 (48.521) | 52.70 (46.015)
  Month 12 (n=35, 41, 40) | 53.58 (47.785) | 53.63 (48.358) | 58.03 (46.264)

17. Secondary Outcome: Percentage of Asthma Symptom Free Days
Description: Days without Asthma Symptom documented in the participant's diary were reported.
Time Frame: Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
percentage of days
  Month 1 (n=62, 60, 60) | 37.32 (40.983) | 36.95 (42.207) | 35.00 (43.032)
  Month 2 (n=61, 50, 56) | 38.47 (44.743) | 41.16 (44.738) | 33.56 (44.161)
  Month 4 (n=54,55, 59) | 42.57 (46.573) | 38.83 (44.042) | 35.78 (43.538)
  Month 6 (n=53, 50, 51) | 41.75 (46.474) | 39.87 (43.744) | 40.09 (45.274)
  Month 8 (n=46, 46, 46) | 38.86 (43.312) | 43.90 (45.377) | 40.03 (43.369)
  Month 10 (n=43, 47, 44) | 41.00 (46.575) | 41.65 (47.435) | 39.83 (44.332)
  Month 12 (n=42, 44, 45) | 43.20 (46.787) | 42.03 (47.093) | 44.61 (46.120)

18. Secondary Outcome: Quality of Life Assessments as Per Paediatric Asthma Quality of Life Questionnaire, Standardized (PAQLQ[S])
Description: The PAQLQ(S) consists of 23 items divided into three domains: Activity limitations (items 1-3, 19, 22); Symptoms (items 4, 6, 8, 10, 12, 14, 16, 18, 20, 23) and Emotional function (items 5, 7, 9, 11, 13, 15, 17, 21). Participants were asked to answer each question using a seven-point scale (where "1" indicated maximum impairment and "7" indicated no impairment) and recall their experience during the previous week. Overall PAQLQ score is equal to the mean of all 23 items for a total possible score 1 (worst) to 7 (best).
Time Frame: Months 2, 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
score on a scale
  Month 2 (n=70, 73, 75) | 6.21 (0.979) | 6.27 (0.878) | 6.08 (1.031)
  Month 6 (n=65, 72, 72) | 6.33 (0.874) | 6.26 (0.982) | 6.30 (0.933)
  Month 12 (n=64, 69, 65) | 6.42 (0.786) | 6.34 (0.946) | 6.36 (0.824)

19. Secondary Outcome: Quality of Life Assessments as Per Paediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ)
Description: The PACQLQ consists of 13 items divided into two domains: Activity limitations (items 2, 4, 6, 8) and Emotional function (items 1, 3, 5, 7, 9, 10, 11, 12, 13). Caregivers answered each question using a seven-point scale (whereby "1" indicated maximum impairment and "7" indicated no impairment) and recalled their experiences during the previous week. Overall PACQLQ score is equal to the mean of all 13 items for a total possible score of 1 (worst) to 7 (best).
Time Frame: Months 2, 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
score on a scale
  Month 2 (n=73, 73, 76) | 5.87 (1.196) | 6.16 (1.033) | 6.08 (1.078)
  Month 6 (n=67, 72, 73) | 6.15 (1.005) | 6.16 (1.115) | 6.31 (0.927)
  Month 12 (n=66, 69, 66) | 6.32 (0.849) | 6.25 (0.712) | 6.31 (0.899)

20. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Findings
Description: Vital signs included body temperature, systolic and diastolic blood pressure and heart rate in beats per minute (bpm). The investigator determined if the result was clinically significant based on the following criteria: Systolic Blood Pressure >130 mmHg or <80 mmHg or a >20 mmHg difference from Baseline; Diastolic Blood Pressure > 85 mmHg; and Resting Heart Rate >140 bpm or <60 bpm or a >30 bpm difference from Baseline.
Time Frame: Up to 12 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
participants | 0 (0) | 0 (0) | 0 (0)

21. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: A thorough physical examination was performed consisting of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) lungs/thorax; (4) heart/cardiovascular system; (5) abdomen; (6) skin and mucosae; (7) nervous system; (8) lymph nodes; (9) musculo-skeletal system; (10) physical examinations other than body systems described in (1) to (9). The investigator determined if any of the findings were clinically significant.
Time Frame: Up to 12 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
participants | 0 (0) | 0 (0) | 0 (0)

22. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Clinically significant laboratory values were hematology and chemistry tests determined by the investigator to be clinically significant based on the following criteria: Hemoglobin <9.5 g/dL; Erythrocytes <3.0 x 10^6/μL or >6.5 x 10^6/μL; White Blood Count <3000/mm^3 or >20000/mm^3; serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), gamma-glutamyl transpeptidase (GGT), Total Bilirubin and Glucose >2 times Upper limit of Normal Range (ULNR); Alkaline Phosphatase and Creatine Kinase >3 times ULNR; Creatinine >1.5 times ULN; Potassium >5.0 mmol/L or <3.0 mmol/L; and Sodium >150 mmol/L or 130 mmol/L.
Time Frame: Up to 12 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
participants | 0 (0) | 0 (0) | 0 (0)

23. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect or any other important medical condition considered serious based on medical and scientific judgement.
Time Frame: Up to 12 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Number analyzed (Participants) | 79 | 76 | 84
participants
  Adverse Events | 61 | 64 | 63
  Serious Adverse Events | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to treatment. All adverse events and serious adverse events were coded according to MedDRA versions 8.0, 8.1, 9.0 and 9.1.
Arm/Group | Ciclesonide 100 µg | Ciclesonide 200 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/79 | 2/76 | 2/84
Other Adverse Events (participants affected / at risk) | 56/79 | 55/76 | 56/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide 100 µg (N=79) | Ciclesonide 200 µg (N=76) | Placebo (N=84)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Myringoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide 100 µg (N=79) | Ciclesonide 200 µg (N=76) | Placebo (N=84)
Pyrexia (General disorders) | 6 (6) | 2 (2) | 4 (5)
Ear infection (Infections and infestations) | 5 (5) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 6 (8) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 13 (20) | 9 (18) | 14 (30)
Pharyngitis (Infections and infestations) | 5 (5) | 4 (5) | 4 (5)
Rhinitis (Infections and infestations) | 4 (4) | 0 (0) | 3 (5)
Sinusitis (Infections and infestations) | 1 (2) | 1 (1) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 18 (28) | 19 (31) | 16 (35)
Headache (Nervous system disorders) | 4 (6) | 7 (10) | 8 (10) — non-serious
Asthma (Respiratory, thoracic and mediastinal disorders) | 35 (60) | 38 (64) | 39 (82) — non-serious
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (10) | 6 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days